CLINICAL TRIAL: NCT00245713
Title: 9-11 Week Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Study to Determine Effects of Adjunctive Levetiracetam on Sleep Architecture of Adults With Partial Onset Epilepsy Receiving a First Generation Anti-epileptic Drug.
Brief Title: Determine Effects of Adjunctive Levetiracetam on Sleep Architecture in Adults With Partial Onset Epilepsy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: N01085
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy, Partial
Keywords: Levetiracetam, adult, partial-onset epilepsy, antiepileptic
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam

INTERVENTIONS:
Drug: levetiracetam

SUMMARY:
Effect of adjunctive levetiracetam on polysomnography in adults with partial-onset epilepsy receiving a classical antiepileptic drug

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have partial onset epilepsy and have been taking carbamazepine or phenytoin at a stable dose for a period of 4 weeks prior to the selection visit
* Subjects must have controlled partial onset seizures which can potentially benefit from adjunctive treatment

Exclusion Criteria:

* Subjects dosing with LEV two weeks prior to the selection visit
* Subjects using more than one AED
* Subjects with specific and non-specific sleep disorders

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Enrollment: 40
Dates: Start 2003-03; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline to visit 7 in percent REM, percent slow wave sleep (stages 3 and 4), and sleep efficiency (which is total sleep time ÷ time in bed defined as lights out), with particular focus on sleep efficiency.

SECONDARY OUTCOMES:
Secondary endpoints are based on the changes from Baseline to visit 7

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma